CLINICAL TRIAL: NCT04510714
Title: A Prospective, Phase III Study to Assess the Efficacy and Safety of Microwave Ablation of Metastatic Lung Sarcoma Lesions.
Brief Title: BORIS - aBlação pOR mIcro-ondaS [Microwave Ablation]
Acronym: BORIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Collaborators: Angiodynamics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 804/15
Record Dates: First submitted 2020-08-10; First posted 2020-08-12 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-02

CONDITIONS: Sarcoma
Keywords: Sarcoma; Percutaneous ablation; Lung ablation; Microwave ablation
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Microwave ablation arm (Experimental): Single arm patients with lung sarcoma metastasis that will be treated with microwave ablation
  Interventions: Device: Image guided percutaneous microwave ablation

INTERVENTIONS:
Device: Image guided percutaneous microwave ablation — Lung metastasis from sarcoma will be treated with microwave antennas (SOLERO) and Ablation System and microwave generators (Angiodynamics), with power settings of 35-45W and an average ablation time of 15 minutes (range 10-30 minutes). The ablation time will be recorded for all procedures. The manufacturer's recommendations will be observed in all cases, since it is assured that patients are able to tolerate the total ablation time.
  Other Names: Image guided percutaneous lung metastasis ablation

SUMMARY:
Patients with sarcoma and lung metastases have few therapeutic options, with poor response to systemic treatment. Many of them are not eligible to surgical treatments due to the high number and distribution of pulmonary lesions or due to comorbidities, which reduce the survival chances of these individuals. Given the high efficacy and overall increased survival demonstrated by recent studies, the minimally invasive treatments (mainly radiofrequency ablation) have gained ground. Although the microwave ablation is a promising new technique for the treatment of patients with pulmonary metastases, there are few studies in the literature to evaluate the efficacy and safety of this procedure in the above population.

DETAILED DESCRIPTION:
This study was designed to prospectively evaluate the safety and effectiveness of microwave ablation therapy in the treatment of metastatic lung lesions secondary to sarcoma. This technique has been proven to be successful in producing greater areas of ablation, increasing the chances of success and reducing the possibility of local recurrence, especially when compared to radiofrequency ablation. There will be 60 consecutive patients diagnosed and treated at the oncology clinic at the São Paulo State Cancer Institute that are going to participate in this study, after meeting the inclusion/ exclusion criteria. This number may be increased up to approximately about 20 patients, according to the sample behavior in the initial analysis and follow-up. All patients will be informed about the benefits, risks, complications and limitations related to the procedure and written informed consent will be applied. Patients will also be informed that microwave ablation is a new technology in Brazil, despite the extensive international experience and the results already validated in the medical literature.

Logistic regression will be used to evaluate the success of the microwave ablation according to the characteristics of the lesion before the procedure. Logistic regressions for correlated data will be used to (a) evaluate the success of ablation according to all registered lesion characteristics, i.e., numeric characteristics (including tumor size and location) and categorical characteristics (histopathology of the primary tumor); (b) verify if combinations of two or more features of the lesions pose significant independent predictors for the success of ablation; and (c) construct a model to estimate the probability of success of the microwave ablation based on lesion characteristics before the procedure. The survival of patients will be assessed according to (a) the end result of the procedure (patients will be classified in two groups: an effective ablation group and a non-effective ablation group) and (b) the histopathological nature of the primary tumor. The survival rates will be calculated using the Kaplan-Meier test. The log-rank test (x² value of Cox-Mantel) will be used to determine statistically significant differences between the patients' survival rates. The value of P less than 0.05 will be considered to indicate a statistically significant difference for all analyses. Statistical software (Bias for Windows, version 8.4, Epsilon Verlag, Frankfurt, Germany) will be used.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years;
* Patients with lung metastases arising from sarcoma;
* Patients who are not eligible for surgery for medical reasons, including limited cardiopulmonary reserve. In this cases we will perform a pulmonary function test (PFT) to determine if the patient can withstand ablation;
* Patients with recurrent metastases after pneumectomy or metastases after surgical resection. In this cases we will perform a PFT to determine if the patient can withstand ablation;
* Patients with pulmonary lesions with dimensions up to 3,0 cm in the largest axial diameter;
* Patients with four or fewer lesions. In cases of bilateral metastases, we will evaluate the treatment of only one lung at a time, with an interval of at least two weeks for the treatment of the contralateral lung, respecting the clinical evolution of the patient.
* Patients with no extrapulmonary metastases or just indolent extrapulmonary disease;
* Patients with prior histopathological confirmation of pulmonary lesions.

Exclusion Criteria:

* Patients with primary disease without clinical control;
* Presence of uncontrolled extrapulmonary disease, including lymph node progression;
* Presence of hilar lesions or near the main bronchi;
* Presence of five or more lung lesions and/or lesions larger than 3,0 cm in greatest axial length;
* Presence of tumors infiltrating the chest wall, mediastinal and/or pleural dissemination;
* Patients with severe coagulopathy (international normalized ratio (INR) > 1,5 or lower platelet count to 50000/mm³);
* Patients with chronic obstructive pulmonary disease (COPD) stage III/ IV;
* Patients with septicemia;
* Patients refusing ablation treatment or participation in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3 years
  Patients with sarcoma pulmonary metastases who are treated with microwave ablation of lung lesions may have higher overall survival rates compared to patients not subject to any kind of treatment or even chemotherapy/ palliative treatment. The literature contains data favorable to treating these patients with microwave ablation, since higher survival rates have been observed, especially when handled all lung lesions (R0).

CONTACTS AND LOCATIONS:
Overall Officials: Marcos Roberto de Menezes, MD, PHD, Principal Investigator — Instituto do Cancer do Estado de Sao Paulo
Locations (1):
- Instituto do Câncer do Estado de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] Vogl TJ, Naguib NN, Gruber-Rouh T, Koitka K, Lehnert T, Nour-Eldin NE. Microwave ablation therapy: clinical utility in treatment of pulmonary metastases. Radiology. 2011 Nov;261(2):643-51. doi: 10.1148/radiol.11101643. PMID 22012906
- [Background] Abbas G, Schuchert MJ, Pennathur A, Gilbert S, Luketich JD. Ablative treatments for lung tumors: radiofrequency ablation, stereotactic radiosurgery, and microwave ablation. Thorac Surg Clin. 2007 May;17(2):261-71. doi: 10.1016/j.thorsurg.2007.03.007. PMID 17626404
- [Background] Dupuy DE, Mayo-Smith WW, Abbott GF, DiPetrillo T. Clinical applications of radio-frequency tumor ablation in the thorax. Radiographics. 2002 Oct;22 Spec No:S259-69. doi: 10.1148/radiographics.22.suppl_1.g02oc03s259. PMID 12376615
- [Background] Wolf FJ, Grand DJ, Machan JT, Dipetrillo TA, Mayo-Smith WW, Dupuy DE. Microwave ablation of lung malignancies: effectiveness, CT findings, and safety in 50 patients. Radiology. 2008 Jun;247(3):871-9. doi: 10.1148/radiol.2473070996. Epub 2008 Mar 27. PMID 18372457
- [Background] Dupuy DE, Zagoria RJ, Akerley W, Mayo-Smith WW, Kavanagh PV, Safran H. Percutaneous radiofrequency ablation of malignancies in the lung. AJR Am J Roentgenol. 2000 Jan;174(1):57-9. doi: 10.2214/ajr.174.1.1740057. No abstract available. PMID 10628454
- [Background] Simon CJ, Dupuy DE, DiPetrillo TA, Safran HP, Grieco CA, Ng T, Mayo-Smith WW. Pulmonary radiofrequency ablation: long-term safety and efficacy in 153 patients. Radiology. 2007 Apr;243(1):268-75. doi: 10.1148/radiol.2431060088. PMID 17392258
- [Background] Suh R, Reckamp K, Zeidler M, Cameron R. Radiofrequency ablation in lung cancer: promising results in safety and efficacy. Oncology (Williston Park). 2005 Oct;19(11 Suppl 4):12-21. PMID 16366374
- [Background] Nakamura T, Matsumine A, Yamakado K, Matsubara T, Takaki H, Nakatsuka A, Takeda K, Abo D, Shimizu T, Uchida A. Lung radiofrequency ablation in patients with pulmonary metastases from musculoskeletal sarcomas [corrected]. Cancer. 2009 Aug 15;115(16):3774-81. doi: 10.1002/cncr.24420. PMID 19514086
- [Background] Ding JH, Chua TC, Glenn D, Morris DL. Feasibility of ablation as an alternative to surgical metastasectomy in patients with unresectable sarcoma pulmonary metastases. Interact Cardiovasc Thorac Surg. 2009 Dec;9(6):1051-3. doi: 10.1510/icvts.2009.218743. Epub 2009 Sep 18. PMID 19767303
- [Background] Lu Q, Cao W, Huang L, Wan Y, Liu T, Cheng Q, Han Y, Li X. CT-guided percutaneous microwave ablation of pulmonary malignancies: Results in 69 cases. World J Surg Oncol. 2012 May 7;10:80. doi: 10.1186/1477-7819-10-80. PMID 22564777